CLINICAL TRIAL: NCT03419715
Title: A Phase IIa Randomized, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Bimatoprost in the Treatment of Migraine
Brief Title: Topical Bimatoprost in the Treatment of Migraine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Manistee Partners (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-MAN-001
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Migraine Disorders; Headache Disorders
Keywords: migraine; headache; bimatoprost
MeSH Terms: conditions — Migraine Disorders; Headache Disorders; Headache | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bimatoprost Topical Solution (Experimental): 0.03% bimatoprost topical solution applied daily to the nail bed of fingers on one hand for 12 weeks
  Interventions: Drug: Bimatoprost Topical Solution
- Control (Placebo Comparator): Saline placebo topically applied daily to the nail be of fingers on one hand for 12 weeks
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Bimatoprost Topical Solution — One drop of bimatoprost topical solution is applied daily to the lunula region of the fingernail bed
  Other Names: Lumigan
  Arms: Bimatoprost Topical Solution
Drug: Control — One drop of saline solution is applied daily to the lunula of the fingernail bed on one hand.
  Other Names: placebo
  Arms: Control

SUMMARY:
The study is to assess the effectiveness of topically applied bimatoprost in reducing migraine headache frequency, severity, and duration. It will also assess the effect of topical bimatoprost on quality of life.

DETAILED DESCRIPTION:
Hall, et al. have observed retrospectively that treatment with topical prostaglandin F2 alpha analogs (applied either to the eye or fingernail bed) significantly reduced the frequency, severity and duration of headaches in migraine sufferers, as well as their migraine disability assessment score (MIDAS).

This is a double-blind, placebo-controlled prospective clinical study to determine if the effect of FDA-approved bimatoprost, a prostaglandin F2 alpha analogue, has anti-migraine activity when administered topically to people suffering from migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraines based on International Classification of Headache Disorders (ICHD) II criteria and experiencing headaches for 4 or more days per month.

Exclusion Criteria:

* Significant liver or renal dysfunction,
* On treatment for inflammatory bowel disease, medication over-use for headaches according to the ICHD II criteria,
* Use of antipsychotics in the past month,
* Recent (in the past six months) history of alcohol or drug abuse,
* Allergy to bimatoprost and its compounds,
* Severe comorbid psychiatric illness,
* Severe infection,
* Malignancy,
* Severe cardiovascular disease,
* Neurodegenerative disorders,
* Pregnancy and lactation, and
* Sexually active women of child bearing age who do not use any method of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in Headache Frequency | 12 weeks
  Change from baseline in the average number of headache days per month

SECONDARY OUTCOMES:
Intensity of Headaches | 12 weeks
  Change from baseline in the average intensity of headaches on a scale of 0 (no pain at all) to 10 (life-threatening pain)
Duration of Headaches | 12 weeks
  Change from baseline in the average duration of headaches
Migraine Disability Assessment Scale (MIDAS)--Quality of Life | 12 weeks
  Change from baseline in quality of life as measured by the Migraine Disability Assessment Scale (MIDAS). MIDAS is a five-item instrument developed to measure migraine related disability and functional consequences. It is divided into four categories based on the score of: 0-5, minimal disability; 6-10, mild disability; 11-20, moderate disability; greater than 20; severe disability.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Bratzler, PhD, Study Chair — Manistee Partners
Locations (2):
- United States (2):
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Omega Medical Research, Warwick, Rhode Island

REFERENCES:
- [Result] Hall LB et al. The Effect of Topical Prostaglandins on Migraine Headaches. Poster Presentation at the Association for Research in Vision and Ophthalmology Annual Meeting, May 2017.

DOCUMENTS (1):
  • Study Protocol (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT03419715/Prot_000.pdf